CLINICAL TRIAL: NCT00113321
Title: Phase II Study of Low-Dose Decitabine (5-AZA-2'-Deoxycytidine) in Myelodysplastic Syndrome (MDS) Post Azacytidine (AZA) Failure
Brief Title: Low-Dose Decitabine in Myelodysplastic Syndrome Post Azacytidine Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0468
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
Keywords: Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia; Azacytidine Failure; Decitabine
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine (Experimental): 20 mg/m2 by vein (IV) over 1 hour daily x 5 days.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 20 mg/m2 IV over 1 hour daily x 5 days.
  Other Names: Dacogen®

SUMMARY:
To study if decitabine can help to control Myelodysplastic Syndrome (MDS) in patients who have failed on therapy with azacytidine, the current standard of therapy.

DETAILED DESCRIPTION:
Methylation is a change that occurs to Deoxyribonucleic acid (DNA) that affects gene usage in human cells. Abnormal methylation is very common in leukemias, which is a related disease to MDS. Decitabine is a new drug that blocks DNA methylation. Researchers want to find out if blocking methylation will help control MDS.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a physical exam, routine blood tests (between 4-6 tablespoons), and a bone marrow aspirate. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

If you are found to be eligible to take part in this study, you will receive decitabine by vein over one hour, once a day, for 5 days (1 course). If this is not possible due to complications, you will receive the drug as an injection under the skin twice a day for 5 days (1 course). Treatment will be given every 4 to 8 weeks depending on how well your blood counts recover.

After completing 8-12 weeks of therapy, response will be evaluated. If the response to treatment is good, treatment with decitabine will continue. Decitabine treatment may be continued for up to 12 courses, or as long as it is judged best to control the leukemia.

During this study, you will need to visit your doctor periodically for physical exams and measurement of vital signs. The frequency of doctor visits will vary depending on your physical condition, but will be required at least once a month.

Blood tests (about 2 teaspoons) will be done about every week during the first 6-8 weeks of treatment, then every 1 to 2 weeks for the length of the study. The blood samples will be used for routine lab tests. Every 1-3 courses, bone marrow samples will also be taken to check cells related to the disease before, during (every 1-3 courses), and after completion of this study.

You will be taken off study if the disease gets worse or intolerable side effects occur.

This is an investigational study. Decitabine is not yet Food and Drug Administration (FDA)approved. It will be provided free of charge by MGI Pharma. Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. MDS and 5% or more marrow blasts, or IPSS risk intermediate 1-2 or high risk; or chronic myelomonocytic leukemia. Patients must have failed therapy with azacytidine.
2. Performance status 0-2 (ECOG scale); adequate hepatic (bilirubin < 2 mg/dl) and renal functions (creatinine <2mg/dl); New York Heart Association (NYHA)cardiac status III-IV excluded.
3. Signed informed consent.
4. No prior intensive combination chemotherapy or high-dose ara-C (>/= 1g/m*2 per dose). Prior biologic therapies, targeted therapies and single agent chemotherapy allowed.
5. Patients must have been off chemotherapy for 2 weeks prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease. Use of hydroxyurea for patients with rapidly proliferative disease is allowed for the first two weeks on therapy.

Exclusion Criteria:

1. Nursing and pregnant females are excluded. Patients of childbearing potential should practice effective methods of contraception. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
2. Patients with active and uncontrolled infections.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Kantarjian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 3/28/05 - 11/7/08; all patients were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Study was terminated due to low accrual.
Period: Overall Study
Arm/Group | Decitabine
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 15
Age Continuous [Median (Full Range); unit: years] | 75 [58 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Participants with Overall Response, categorized as 'Complete Response' to represent remission or 'No Complete Response' for lack of remission. Response evaluation after completing one course of therapy (8-12 weeks), then bone marrow aspiration to document remission every 1-3 courses.
Time Frame: Blood tests baseline and after completing 8-12 weeks of therapy
Population: Treated population (16 patients); No further analysis done since study terminated early due to low accrual.
Measure: Number; unit: Participants
Arm/Group | Decitabine
Number analyzed (Participants) | 16
Participants
  Complete Response | 3
  No Complete Response | 13

ADVERSE EVENTS:
Time Frame: 2 years 1 month
Arm/Group | Decitabine
Serious Adverse Events (participants affected / at risk) | 6/16
Other Adverse Events (participants affected / at risk) | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=16)
Death (General disorders) | 3 (3)
Febrile Neutropenia (Infections and infestations) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated to study drug.
Elevated Cardiac Triponin (Cardiac disorders) | 1 (1)
Blood/Bone Marrow (Other) - Spleen (Blood and lymphatic system disorders) | 1 (1) — Patient had history of splenomegaly
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=16)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated Alanine transaminase (ALT) (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 7 (7)
Elevated aspartate aminotransferase (AST) (Metabolism and nutrition disorders) | 7 (7)
Elevated Bilirubin (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Elevated Creatinine (Metabolism and nutrition disorders) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Metabolic/Laboratory (0ther) (Metabolism and nutrition disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Pain (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No